CLINICAL TRIAL: NCT07227259
Title: Assessment of Systematic Health Properties of Pecan Nut Consumption: Gut, Vascular, Metabolic and Cognitive Outcomes
Brief Title: Health Properties of Pecan Nut Consumption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Francene Steinberg, Professor, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2340870
Record Dates: First submitted 2025-11-09; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adults
Keywords: pecan nut; cardiovascular; gut microbiome; cognitive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecan nut then no nut (Experimental): Participant will add pecan nuts to their diet during the first intervention arm, then they will cross over to the no nut diet arm
  Interventions: Other: pecan nut
- No nut then pecan nut (Experimental): Participant will consume a diet without nuts during the first intervention arm, then they will cross over to the arm where they will add pecan nuts to their diet.
  Interventions: Other: pecan nut

INTERVENTIONS:
Other: pecan nut — Dose - 2 ounces of pecan nuts, daily

SUMMARY:
The main goal of this clinical study is to see if consuming pecan nuts will result in improvements in overall body metabolism such as in blood lipids, markers of inflammation, blood pressure, cognitive performance and changes in bacteria living in the gut in adults 45 to 75 years of age.

Participants will take part in two 3-month intervention periods, separated by 4-6 weeks, in random order ( a total of approximately 7 months). During one intervention period, they will include pecan nuts in their diet each day, while during the other intervention period they will avoid pecans in their diet. There will be an initial screening visit to evaluate eligibility and four study visits to the clinic.

Participants will be asked to complete some questionnaires about their diet, physical and cognitive health, and provide blood and stool samples, and have their blood pressure measured.

ELIGIBILITY:
Inclusion Criteria: BMI of 20-35 kg/m2, ability to understand the intervention instructions, Willingness to follow the dietary intervention, willingness to provide biological samples (blood and stool) -

Exclusion Criteria: allergy to pecan or other nuts, cognitive impairment due to dementia of any type and inability to understand or comply with intervention instructions, use of menopausal hormone replacement therapy, use of antibiotics or probiotics in the 2 months prior to enrollment, uncontrolled diabetes with HbA1C of >9.5, vegetarian/vegan, any serious medical condition (such as chronic kidney disease of stage 3 or greater, heart failure, active cancer treatment, inflammatory bowel disease, etc.), consumption of supplements that may interfere with vascular response or gut microbiome, use of statin drugs for cholesterol lowering.

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in vascular response at 3 months | Change from baseline at 3 months
  Vascular response as measured by Pulse Wave Velocity (PWV)

SECONDARY OUTCOMES:
Change in blood lipids over 3 months | Change from baseline at 3 months
  Blood lipids as measured by clinical lipid panel, including total, LDL and HDL cholesterol, and Tiglycerides
Change in markers of inflammation at 3 months | change from baseline at 3 months
  Markers of inflammation as measured by Luminex cytokine panel IL-17
Change in gut microbiome profile at 3 months | Change from baseline at 3 months
  Gut microbiome profile as measured by fecal 16S rRNA gene sequencing
Change in blood markers of intestinal permeability at 3 months. | Change from baseline at 3 months
  Blood marker of intestinal permeability as measured by ELISA for LBP and LPS
Change in blood markers of intestinal permeability at 3 months | Change from baseline at 3 months
  Blood biomarker of intestinal permeability and immune activation as measured by ELISA of sCD14
Change in cognitive function - reaction time at 3 months | Change from baseline at 3 months
  Reaction time task as measured by CANTAB assessments
Change in cognitive function - working memory at 3 months | Change from baseline at 3 months
  Spatial working memory as assessed by CANTAB
Change in cognitive function - episodic memory at 3 months | Change from baseline to 3 months
  Paired associates learning as measured by CANTAB
Change in cognitive function - sustained attention at 3 months | Change from baseline at 3 months
  Attention measured via Rapid visual information processing using CANTAB
Change in quality of life at 3 months | Change from baseline at 3 months
  Self-perceived quality of life questionnaire assessed using World Health Organization Qualigy of Life Instruments (WHOQOL-BREF)
Change in sleep quality at 3 months | Change from baseline at 3 months
  Self-rated questionnaire of sleep quality measured by Pittsburgh Sleep Quality Index (PSQI)
Change in mood over 3 months | Change from baseline to 3 months
  Assessment of mood using the Affect Grid
Change in perceived stress over 3 months | Change from baseline at 3 months
  Assessment of stress using the Perceived Stress Scale (PSS-10)
Change in anxiety at 3 months | Change from baseline at 3 months
  Anxiety measured using the Generalized Anxiety disorder Scale (GAD-7)
Change in depressive symptoms at 3 months | Change from baseline at 3 months
  Assessment of depressive symptoms using the Beck Depression Inventory-II (BDI-II)
Change in blood acute phase inflammatory response maker at 3 months | Change from baseline at 3 months
  Acute phase inflammatory response measured by hsCRP

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Center, UC Davis campus, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No